CLINICAL TRIAL: NCT03849807
Title: The Effects of Chiropractic Care on Behavior, Neurological Function and Quality of Life in Children With Attention Deficit Hyperactivity Disorder: A Randomized Controlled Pilot Study
Brief Title: Chiropractic Care on Behavior, Neurological Function and Quality of Life in ADHD Children - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Imran khan Niazi2
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; Children; Chiropractic; Neurological function; Quality of life
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Successful blinding of patients or practitioners in a trial involving a physical intervention such as chiropractic care is virtually impossible.18 This is due to the manual nature of the interventions and the challenges associated with providing appropriate sham procedures.18, 19 However, participants in this trial are highly likely to be naïve to chiropractic care so it is possible they will remain unaware of whether they are in the chiropractic or control group. Some study personnel will be aware of the allocated arm as they will be responsible for logistical aspects of the trial. However, the research specialist collecting and analyzing data during the trial will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Chiropractic care
  Interventions: Other: Experimental group
- Control group (Active Comparator): Usual health care
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — the intervention group will receive 4 weeks of chiropractic care along with usual care(Cognitive-Behavioral, psychosocial Therapy).
  Arms: Experimental group
Other: Control group — Participants in the group will receive usual health (Cognitive-Behavioral, psychosocial Therapy) care or wish to engage in during the course of the study as well as receiving a passive movement control intervention delivered by a chiropractor 3 times per week in the same hospital setting as the group receiving chiropractic care.
  Arms: Control group

SUMMARY:
To date the effects of chiropractic care on behavior and neurological function in children diagnosed with ADHD has not been investigated thoroughly and is limited mostly to case studies and retrospective case reviews. Our research group recently completed a pilot study that investigated the effects of a single session of chiropractic care on oculomotor function and reading ability in children with ADHD. The findings of this study suggested that chiropractic care may have a role in improving oculomotor control and reading ability in this population group. This proposed study is the next step in this program of research and is a pilot clinical trial that will investigate whether 4 weeks of chiropractic care influences behavior, neurological function, or quality of life in children with ADHD.

DETAILED DESCRIPTION:
ADHD is a disorder that may affect an individual's academic performance, social interactions, and interpersonal relationships amongst others. It is characterized by impulsiveness, hyperactivity, and inattention. It was previously thought that children overcome ADHD as they grow up, however, recent studies suggest that 30-60% of affected individuals continue to show significant symptoms of the disorder as adults and have associated difficulties such as lower educational and employment achievement. Conventional therapeutic approaches that are used with individuals with ADHD generally involve pharmaceutical interventions and behavioral therapies such as counseling and behavioral modification. However, little is known about the long term effectiveness of these treatment approaches which are also known to involve significant risks and complications.

ADHD is a neurodevelopmental disorder that is associated with significant alterations in brain development and function. These include changes in fronto-striatal pathways that can lead to difficulties with "top-down" control. It is also likely that connections in the parietal lobe and cerebellum are involved. These neurological changes are associated with a number of alterations to sensory filtering, sensorimotor gating, and sensorimotor control. This lends itself to a potential role for chiropractors in caring for children with ADHD because chiropractic care has been shown to alter a number of aspects of sensorimotor function.

Chiropractic is based on the theory that spinal adjustments applied to areas of spinal dysfunction, known as vertebral subluxations, can improve the function of the nervous system. Our research group has been testing this theory for the last 15 years. We have hypothesized that the articular dysfunction component of the vertebral subluxation results in altered afferent input to the central nervous system (CNS) that modifies the way in which the CNS processes and integrates all subsequent sensory input. This processing (i.e. sensorimotor integration), is a CNS function that appears most vulnerable to altered inputs. Recent studies have shown that chiropractic care alters sensorimotor filtering, cortical and cerebellar motor processing, and multisensory processing, all of which may be important in the neurodevelopment of ADHD. Given the nature of the neurological changes associated with ADHD and the growing body of evidence that suggests that chiropractic care may influence neurological function, it is possible that chiropractors may play a role in enhancing the neurological function of individuals with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* have been previously diagnosed with Attention Deficit Hypersensitivity Disorder based on the criteria outlined in the DSM-V.

Exclusion Criteria:

* have absolute contraindications to chiropractic adjustments
* have experienced previous significant adverse reactions to chiropractic care or manual therapies.
* investigators are unable to get consent from parents and caregivers of participating children in the trial

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Vanderbilt Attention Deficit Hyperactivity Disorder (ADHD) Diagnostic Rating Scale | baseline,4th week, 8th week
  Changes From Baseline, The Vanderbilt ADHD Diagnostic Rating Scale (VADRS) is a psychological assessment tool for Attention Deficit Hyperactivity Disorder (ADHD) symptoms and their effects on behavior and academic performance in children. It have two components: symptom assessment and impairment in performance. To meet criteria for ADHD diagnoses, one must have 6 positive responses to either the core 9 inattentive symptoms or core 9 hyperactive symptoms, or both. the respondent to rate the frequency of a child's behaviors on a 0-3 scale as follows: 0: "never"; 1: "occasionally"; 2: "often"; 3: "very often".
  to rate the child's performance in school and his or her interactions with others on a 1-5 scale, with 1-2 meaning "above average", 3 meaning "average", and 4-5 meaning "problematic". To meet criteria for ADHD, there must be at least one score for the performance set that is either a 4 or 5, as these scores indicate impairment in performance.
Swanson, Nolan and Pelham (SNAP) Questionnaire | baseline,4th week, 8th week
  Changes from the Baseline The SNAP-IV is based on a 0 to 3 rating scale: Not at All = 0, Just A Little = 1, Quite A Bit = 2, and Very Much = 3. Subscale scores on the SNAP-IV are calculated by summing the scores on the items in the subset and dividing by the number of items in the subset.
ADHA Attention Deficit Hyperactivity Disorder Rating Scale IV (Home version) | baseline,4th week, 8th week
  Changes from the Baseline, The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). For inattention (IA) subscale raw score: Add the odd-numbered items
  For hyperactivity-impulsivity (HI) subscale raw score: Add the even-numbered items. To obtain the total raw score: Add the IA and Hi subscale raw scores

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harpin VA. The effect of ADHD on the life of an individual, their family, and community from preschool to adult life. Arch Dis Child. 2005 Feb;90 Suppl 1(Suppl 1):i2-7. doi: 10.1136/adc.2004.059006. PMID 15665153
- [Background] Munoz DP, Armstrong IT, Hampton KA, Moore KD. Altered control of visual fixation and saccadic eye movements in attention-deficit hyperactivity disorder. J Neurophysiol. 2003 Jul;90(1):503-14. doi: 10.1152/jn.00192.2003. Epub 2003 Apr 2. PMID 12672781
- [Background] Sable JJ, Kyle MR, Knopf KL, Schully LT, Brooks MM, Parry KH, Diamond RE, Flink LA, Stowe R, Suna E, Thompson IA. The Sensory Gating Inventory as a potential diagnostic tool for attention-deficit hyperactivity disorder. Atten Defic Hyperact Disord. 2012 Sep;4(3):141-4. doi: 10.1007/s12402-012-0079-1. Epub 2012 May 27. PMID 22644992
- [Background] Haavik H, Murphy B. The role of spinal manipulation in addressing disordered sensorimotor integration and altered motor control. J Electromyogr Kinesiol. 2012 Oct;22(5):768-76. doi: 10.1016/j.jelekin.2012.02.012. Epub 2012 Apr 6. PMID 22483612
- [Background] Henderson CN. The basis for spinal manipulation: chiropractic perspective of indications and theory. J Electromyogr Kinesiol. 2012 Oct;22(5):632-42. doi: 10.1016/j.jelekin.2012.03.008. Epub 2012 Apr 17. PMID 22513367
- [Background] Daligadu J, Haavik H, Yielder PC, Baarbe J, Murphy B. Alterations in cortical and cerebellar motor processing in subclinical neck pain patients following spinal manipulation. J Manipulative Physiol Ther. 2013 Oct;36(8):527-37. doi: 10.1016/j.jmpt.2013.08.003. Epub 2013 Sep 12. PMID 24035521
- [Background] Holt KR, Haavik H, Lee AC, Murphy B, Elley CR. Effectiveness of Chiropractic Care to Improve Sensorimotor Function Associated With Falls Risk in Older People: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2016 May;39(4):267-78. doi: 10.1016/j.jmpt.2016.02.003. Epub 2016 Apr 2. PMID 27050038
- [Background] Karpouzis F, Bonello R, Pollard H. Chiropractic care for paediatric and adolescent Attention-Deficit/Hyperactivity Disorder: A systematic review. Chiropr Osteopat. 2010 Jun 2;18:13. doi: 10.1186/1746-1340-18-13. PMID 20525195
- [Background] Rabe-Jablonska J. [Affective disorders in the fourth edition of the classification of mental disorders prepared by the American Psychiatric Association -- diagnostic and statistical manual of mental disorders]. Psychiatr Pol. 1993 May-Jun;27(3):269-79. No abstract available. Polish. PMID 8356173
- [Background] McGough JJ, Loo SK, Sturm A, Cowen J, Leuchter AF, Cook IA. An eight-week, open-trial, pilot feasibility study of trigeminal nerve stimulation in youth with attention-deficit/hyperactivity disorder. Brain Stimul. 2015 Mar-Apr;8(2):299-304. doi: 10.1016/j.brs.2014.11.013. Epub 2014 Nov 28. PMID 25533244
- [Background] Conners CK. Rating scales in attention-deficit/hyperactivity disorder: use in assessment and treatment monitoring. J Clin Psychiatry. 1998;59 Suppl 7:24-30. PMID 9680050
- [Background] Childress AC, Cutler AJ, Saylor K, Gasior M, Hamdani M, Ferreira-Cornwell MC, Findling RL. Participant-perceived quality of life in a long-term, open-label trial of lisdexamfetamine dimesylate in adolescents with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2014 May;24(4):210-7. doi: 10.1089/cap.2013.0077. Epub 2014 May 9. PMID 24815910
- [Background] Rosner AL. Evidence-based medicine: revisiting the pyramid of priorities. J Bodyw Mov Ther. 2012 Jan;16(1):42-9. doi: 10.1016/j.jbmt.2011.05.003. Epub 2011 Jun 24. PMID 22196426
- [Background] Hancock MJ, Maher CG, Latimer J, McAuley JH. Selecting an appropriate placebo for a trial of spinal manipulative therapy. Aust J Physiother. 2006;52(2):135-8. doi: 10.1016/s0004-9514(06)70049-6. PMID 16764551